CLINICAL TRIAL: NCT01621061
Title: Sleep Apnea and High Altitude Pulmonary Hypertension in Kyrgyz Highlanders
Brief Title: Sleep Related Breathing Disturbances and High Altitude Pulmonary Hypertension in Kyrgyz Highlanders
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Principal Investigator, Konrad E. Bloch, Professor, University of Zurich
Other Study IDs: 01-7/219
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: High Altitude Pulmonary Hypertension; Sleep Apnea
Keywords: high altitude illness; pulmonary hypertension; sleep apnea; hypoxia
MeSH Terms: conditions — Pulmonary edema of mountaineers; Sleep Apnea Syndromes; Hypertension, Pulmonary; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High altitude pulmonary hypertension: Highlanders with high altitude pulmonary hypertension
- High altitude control: Healthy highlanders
- Low altitude control: Healthy lowlanders

SUMMARY:
High altitude pulmonary hypertension, a form of altitude illness that occurs in long-term residents at altitudes >2500 m, is characterized by dyspnea, hypoxemia, impaired exercise performance and hypertension in the pulmonary circulation. Whether sleep related breathing disturbances, common causes of nocturnal hypoxemia in lowlanders, are also prevalent in highlanders and promote pulmonary hypertension in highlanders is unknown. Therefore, the current study will investigate whether highlanders with high altitude pulmonary hypertension have a greater prevalence of sleep apnea than healthy highlanders and lowlanders.

ELIGIBILITY:
Inclusion Criteria:

* high altitude pulmonary hypertension confirmed by clinical presentation and systolic pulmonary artery pressure >50 mmHg measured by echocardiography at altitude of residence.
* healthy subjects (high altitude controls)
* Both genders
* Age >16 y
* Kyrgyz ethnicity
* born, raised and currently living at >2500 m
* healthy subjects currently living at <1000 m (low altitude controls)

Exclusion criteria:

* Pulmonary hypertension from other causes, in particular from left ventricular failure as judged clinically and by echocardiography
* excessive erythrocytosis
* other coexistent disorders that may interfere with the cardio-respiratory system and sleep
* regular use of medication that affects control of breathing
* heavy smoking

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Highlanders with high altitude pumonary hypertension living at an altitude of 2500-4000 m; healthy highlanders living at an altitude of 2500-4000 m; healthy lowlanders living at an altitude of <1000 m.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sleep related breathing disturbances | 4 months
  Nocturnal oxygen saturation and apnea/hypopnea index

SECONDARY OUTCOMES:
Pulmonary artery pressure | 4 months
  Echocardiography
Dyspnea | 4 months
  NYHA functional class
Vigilance | 4 months
  Psychomotor vigilance
Exercise performance | 4 months
  6 min walk test
Pulmonary function | 4 months
  Spirometry
Cerebral oxygen saturation | 4 months
  Near-infrared spectroscopy
Mountain sickness | 4 months
  Quinghai chronic mountain sickness score
Generic quality of life | 4 months
  SF-36 quality of life questionnaire
Disease specific quality of life | 4 months
  Kansas City Cardiomyopathy questionnaire
Subjective sleepiness | 4 months
  Epworth sleepiness scale

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Principal Investigator — University of Zurich, Switzerland; Talant Sooronbaev, MD, Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan